CLINICAL TRIAL: NCT03419182
Title: Randomized Controlled Trial to Determine the Best Treatment of Acetabular Fractures in Geriatric Patients: Open Reduction Internal Fixation With or Without Primary Total Hip Arthroplasty
Brief Title: RCT Determining Best Treatment for Geriatric Acetabular Fractures
Acronym: GeriTab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Theodore Manson, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00047655
Record Dates: First submitted 2017-09-22; First posted 2018-02-01 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Acetabular Fracture
Keywords: Geriatric; Acetabular; Arthroplasty

STUDY DESIGN:
Intervention Model Description: Patients will be randomized t wo treatment groups : 1. Open reduction internal fixation (ORIF) 2. Acute primary total hip athroplasty (THA) +ORIF. These are both two standard accepted treatments for this injury. Participants who do not consent to being randomized will be asked if they would consent to participating in an observational arm. In this case, type of surgery would be planned and chosen by clinical decision making from the surgeon and patient. As these procedures are both standard of care, partipants could end up in either group as well. All follow up will be the same.
Who Masked: Outcomes Assessor
Masking Description: The individual administering the WOMAC or SF-36 will be blinded to the patient's treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RCT - ORIF (Active Comparator): A patient in this study arm consents to randomization and receives RCT - ORIF as his/her treatment assignment. He/she will have his/her acetabular fracture treated by open reduction internal fixation.
  Interventions: Procedure: Open Reduction internal Fixation
- RCT - (THA) + ORIF (Active Comparator): A patient in this study arm consents to randomization and receives RCT - (THA) + ORIF as his/her treatment assignment. He/she will have his/her acetabular fracture treated by open reduction internal fixation with primary total hip arthroplasty.
  Interventions: Procedure: Open Reduction Internal Fixation with Total Hip Arthroscopy
- OBS - ORIF (No Intervention): A patient in this study arm does not consent to randomization, but does agree to be involved in the observational study. He/she decides, with input from his/her surgeon, to have his/her acetabular fracture treated by open reduction internal fixation.
- OBS (THA) + ORIF (No Intervention): A patient in this study arm does not consent to randomization, but does agree to be involved in the observational study. He/she decides, with input from his/her surgeon, to have his/her acetabular fracture treated by open reduction internal fixation with primary total hip arthroplasty.

INTERVENTIONS:
Procedure: Open Reduction internal Fixation — A surgeon uses hardware, such as plates and screws, to restore structural integrity and alignment of an acetabular fracture.
  Arms: RCT - ORIF
Procedure: Open Reduction Internal Fixation with Total Hip Arthroscopy — A surgeon uses hardware, such as plates and screws, to restore structural integrity and alignment of an acetabular fracture, and replaces the cartilage and bone of the greater trochanter with prosthetic components.
  Arms: RCT - (THA) + ORIF

SUMMARY:
There is debate over the best management for acetabular (hip) fractures that occur within the geriatric population. Geriatric patients, 60 years or older, are at greater risk for operative complications because they tend to have poorer bone quality, complicated fractures, and multiple health problems. Physicians currently have no guidelines as to the best surgical management for these particular fractures, because there is little data on the long-term outcomes of these injuries. The use of internal fixation (a nail or plate) is a standard method for repairing these injuries, however when the injuries are complicated it is predicted to have a poorer outcome than performing internal fixation along with total hip arthroplasty (joint reconstruction). Given the significant problems that result from hip fractures in this population, our study is designed to determine the best method for treatment of acetabular fractures and to clarify the criteria for treatment with guidelines assisting the physician in selecting the appropriate treatment.

DETAILED DESCRIPTION:
This is a pilot randomized controlled study conducted at Shock Trauma and University of Maryland Medical Center of patients 60 years and older who have sustained an acetabular fracture. Based on the patient's fracture pattern, dome impaction, posterior wall component and femoral head fracture, the patients will be randomized to their treatment arm. One treatment arm will consist of patients who are treated with ORIF alone. The other treatment will undergo ORIF as well as concomitant total hip arthroplasty in the same surgery.

Furthermore the functional status evaluation of each patient will be standardized using the WOMAC (Western Ontario McMaster Universities OA index), a lower extremity specific outcome score that has been validated for use in patients of similar age to our cohort study in osteoarthritis or after total hip arthroplasty; and the SF-36 (Short Form-36) which is a validated general health outcome measure that calculates mental and physical subcomponent scores. Patients will also be assessed using the Harris Hip Score, which has been used for patients with post-traumatic arthritis undergoing conversion to total hip arthroplasty.

All patients will be followed as standard of care for their follow up visits at 6 month and 1 year. As the patient population at Shock Trauma and University of Maryland Medical Center are all treated by the same orthopaedic group, one dedicated investigator will follow their outcomes. To minimize the risk of bias, I, the individual administering the WOMAC or SF-36 will be blinded to the patient's treatment arm. As the patient will be giving consent for their treatment, they cannot be blinded. Also, the surgeons (and the research coordinator) will know which group the patient is in, but the investigator collecting the data will not.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years and older at the time of injury who have sustained an acetabular fracture
* Fluent in the English Language

Exclusion Criteria:

* Patients under the Age of 60 years old
* Patients who are medically contraindicated for surgery
* Patients who in the surgeon's view will be unable to comply with posterior hip precautions (to prevent dislocation) after surgery
* In patients with bilateral acetabular fractures, the most severe side will be randomized into the study while the other side will be treated but not included in the study.
* Open Injuries

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-04-13 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for this study is the proportion of complications in the first 12 months following surgery | 1 year
  Researchers will assess treatment success using a two-group comparison of proportion of complications between the treatment groups during the first 12 months following treatment.
  Complications will be identified by radiographic and clinical evaluation during standard follow-up appointments with the treating surgeon. Complications include postoperative infections, non-union, mal-union, development of heterotopic bone, development of osteoarthritis, osteolysis, hardware failure, hip dislocations, surgical revisions, and any other condition related to surgical treatment of the study injury.

SECONDARY OUTCOMES:
A secondary outcome for this study is to evaluate patient reported outcomes using the WOMAC Questionnaire. | 6 months and 12 months
  All enrolled patients complete WOMAC questionnaire 6 and 12 months after surgical treatment. Patient reported outcomes are based on scores on the WOMAC questionnaire. Using a mean of 50 and a standard deviation of 10, this study will have 80% power to detect a 10% change in the patient satisfaction questionnaire.
A secondary outcome for this study is to evaluate patient reported outcomes using the SF36 Questionnaire. | 6 months and 12 months
  All enrolled patients complete SF36 questionnaire 6 and 12 months after surgical treatment. Patient reported outcomes are based on scores on the SF36 questionnaire. Using a mean of 50 and a standard deviation of 10, this study will have 80% power to detect a 10% change in the patient satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Manson, MD, Principal Investigator — Associate Professor of Orthopaedics
Locations (1):
- University of Maryland Department of Orthopaedics, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anglen JO, Burd TA, Hendricks KJ, Harrison P. The "Gull Sign": a harbinger of failure for internal fixation of geriatric acetabular fractures. J Orthop Trauma. 2003 Oct;17(9):625-34. doi: 10.1097/00005131-200310000-00005. PMID 14574190
- [Background] Study to Prospectively Evaluate Reamed Intramedullary Nails in Patients with Tibial Fractures Investigators; Bhandari M, Guyatt G, Tornetta P 3rd, Schemitsch EH, Swiontkowski M, Sanders D, Walter SD. Randomized trial of reamed and unreamed intramedullary nailing of tibial shaft fractures. J Bone Joint Surg Am. 2008 Dec;90(12):2567-78. doi: 10.2106/JBJS.G.01694. PMID 19047701
- [Background] Boraiah S, Ragsdale M, Achor T, Zelicof S, Asprinio DE. Open reduction internal fixation and primary total hip arthroplasty of selected acetabular fractures. J Orthop Trauma. 2009 Apr;23(4):243-8. doi: 10.1097/BOT.0b013e3181923fb8. PMID 19318866
- [Background] Buckley R, Tough S, McCormack R, Pate G, Leighton R, Petrie D, Galpin R. Operative compared with nonoperative treatment of displaced intra-articular calcaneal fractures: a prospective, randomized, controlled multicenter trial. J Bone Joint Surg Am. 2002 Oct;84(10):1733-44. doi: 10.2106/00004623-200210000-00001. PMID 12377902
- [Background] Cornell CN. Management of acetabular fractures in the elderly patient. HSS J. 2005 Sep;1(1):25-30. doi: 10.1007/s11420-005-0101-7. PMID 18751805
- [Background] Helfet DL, Borrelli J Jr, DiPasquale T, Sanders R. Stabilization of acetabular fractures in elderly patients. J Bone Joint Surg Am. 1992 Jun;74(5):753-65. PMID 1624491
- [Background] Herscovici D Jr, Lindvall E, Bolhofner B, Scaduto JM. The combined hip procedure: open reduction internal fixation combined with total hip arthroplasty for the management of acetabular fractures in the elderly. J Orthop Trauma. 2010 May;24(5):291-6. doi: 10.1097/BOT.0b013e3181b1d22a. PMID 20418734
- [Background] Jimenez ML, Tile M, Schenk RS. Total hip replacement after acetabular fracture. Orthop Clin North Am. 1997 Jul;28(3):435-46. doi: 10.1016/s0030-5898(05)70300-x. PMID 9208835
- [Background] Kirkley A, Birmingham TB, Litchfield RB, Giffin JR, Willits KR, Wong CJ, Feagan BG, Donner A, Griffin SH, D'Ascanio LM, Pope JE, Fowler PJ. A randomized trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2008 Sep 11;359(11):1097-107. doi: 10.1056/NEJMoa0708333. PMID 18784099
- [Background] Mears DC, Velyvis JH. Acute total hip arthroplasty for selected displaced acetabular fractures: two to twelve-year results. J Bone Joint Surg Am. 2002 Jan;84(1):1-9. doi: 10.2106/00004623-200201000-00001. PMID 11792772
- [Background] Matta JM. Fractures of the acetabulum: accuracy of reduction and clinical results in patients managed operatively within three weeks after the injury. J Bone Joint Surg Am. 1996 Nov;78(11):1632-45. PMID 8934477
- [Background] Moseley JB, O'Malley K, Petersen NJ, Menke TJ, Brody BA, Kuykendall DH, Hollingsworth JC, Ashton CM, Wray NP. A controlled trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2002 Jul 11;347(2):81-8. doi: 10.1056/NEJMoa013259. PMID 12110735
- [Background] Mouhsine E, Garofalo R, Borens O, Fischer JF, Crevoisier X, Pelet S, Blanc CH, Leyvraz PF. Acute total hip arthroplasty for acetabular fractures in the elderly: 11 patients followed for 2 years. Acta Orthop Scand. 2002 Dec;73(6):615-8. doi: 10.1080/000164702321039552. PMID 12553506
- [Background] Osgood GM, Manson TT, O'Toole RV, Turen CH. Combined pelvic ring disruption and acetabular fracture: associated injury patterns in 40 patients. J Orthop Trauma. 2013 May;27(5):243-7. doi: 10.1097/BOT.0b013e31826c2751. PMID 22874118
- [Background] O'Toole RV, Castillo RC, Pollak AN, MacKenzie EJ, Bosse MJ; LEAP Study Group. Determinants of patient satisfaction after severe lower-extremity injuries. J Bone Joint Surg Am. 2008 Jun;90(6):1206-11. doi: 10.2106/JBJS.G.00492. PMID 18519312
- [Background] O'Toole RV, Hui E, Chandra A, Nascone JW. How often does open reduction and internal fixation of geriatric acetabular fractures lead to hip arthroplasty? J Orthop Trauma. 2014 Mar;28(3):148-53. doi: 10.1097/BOT.0b013e31829c739a. PMID 23719343
- [Background] Pellicci PM, Bostrom M, Poss R. Posterior approach to total hip replacement using enhanced posterior soft tissue repair. Clin Orthop Relat Res. 1998 Oct;(355):224-8. doi: 10.1097/00003086-199810000-00023. PMID 9917607
- [Background] Ranawat A, Zelken J, Helfet D, Buly R. Total hip arthroplasty for posttraumatic arthritis after acetabular fracture. J Arthroplasty. 2009 Aug;24(5):759-67. doi: 10.1016/j.arth.2008.04.004. Epub 2008 Jun 4. PMID 18534534
- [Background] Romness DW, Lewallen DG. Total hip arthroplasty after fracture of the acetabulum. Long-term results. J Bone Joint Surg Br. 1990 Sep;72(5):761-4. doi: 10.1302/0301-620X.72B5.2211750.
- [Background] Schulman JE, O'Toole RV, Castillo RC, Manson T, Sciadini MF, Whitney A, Pollak AN, Nascone JW. Pelvic ring fractures are an independent risk factor for death after blunt trauma. J Trauma. 2010 Apr;68(4):930-4. doi: 10.1097/TA.0b013e3181cb49d1. PMID 20386286
- [Background] Stauffer RN. Ten-year follow-up study of total hip replacement. J Bone Joint Surg Am. 1982 Sep;64(7):983-90. PMID 7118986
- [Background] Spencer RF. Acetabular fractures in older patients. J Bone Joint Surg Br. 1989 Nov;71(5):774-6. doi: 10.1302/0301-620X.71B5.2584245.
- [Background] Toro JB, Hierholzer C, Helfet DL. Acetabular fractures in the elderly. Bull Hosp Jt Dis. 2004;62(1-2):53-7. No abstract available. PMID 15517858
- [Background] Weber M, Berry DJ, Harmsen WS. Total hip arthroplasty after operative treatment of an acetabular fracture. J Bone Joint Surg Am. 1998 Sep;80(9):1295-305. doi: 10.2106/00004623-199809000-00008. PMID 9759814
- [Background] Weinstein JN, Lurie JD, Tosteson TD, Skinner JS, Hanscom B, Tosteson AN, Herkowitz H, Fischgrund J, Cammisa FP, Albert T, Deyo RA. Surgical vs nonoperative treatment for lumbar disk herniation: the Spine Patient Outcomes Research Trial (SPORT) observational cohort. JAMA. 2006 Nov 22;296(20):2451-9. doi: 10.1001/jama.296.20.2451. PMID 17119141
- [Background] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Blood E, Hanscom B, Herkowitz H, Cammisa F, Albert T, Boden SD, Hilibrand A, Goldberg H, Berven S, An H; SPORT Investigators. Surgical versus nonsurgical therapy for lumbar spinal stenosis. N Engl J Med. 2008 Feb 21;358(8):794-810. doi: 10.1056/NEJMoa0707136. PMID 18287602
- [Background] Weinstein JN, Lurie JD, Tosteson TD, Hanscom B, Tosteson AN, Blood EA, Birkmeyer NJ, Hilibrand AS, Herkowitz H, Cammisa FP, Albert TJ, Emery SE, Lenke LG, Abdu WA, Longley M, Errico TJ, Hu SS. Surgical versus nonsurgical treatment for lumbar degenerative spondylolisthesis. N Engl J Med. 2007 May 31;356(22):2257-70. doi: 10.1056/NEJMoa070302. PMID 17538085
- [Background] Walley KC, Appleton PT, Rodriguez EK. Comparison of outcomes of operative versus non-operative treatment of acetabular fractures in the elderly and severely comorbid patient. Eur J Orthop Surg Traumatol. 2017 Jul;27(5):689-694. doi: 10.1007/s00590-017-1949-1. Epub 2017 Apr 7. PMID 28389758
- [Background] Shah SB, Manson TT, Nascone JW, Sciadini MF, O'Toole RV. Radiographic Determinants of Early Failure After Posterior Wall Acetabular Fracture Fixation. Orthopedics. 2016 Nov 1;39(6):e1104-e1111. doi: 10.3928/01477447-20160819-03. Epub 2016 Aug 30. PMID 27575037
- [Background] Sterling RS, Krushinski EM, Pellegrini VD Jr. THA after acetabular fracture fixation: is frozen section necessary? Clin Orthop Relat Res. 2011 Feb;469(2):547-51. doi: 10.1007/s11999-010-1612-1. PMID 20945123
- [Background] Manson TT, Perdue PW, Pollak AN, O'Toole RV. Embolization of pelvic arterial injury is a risk factor for deep infection after acetabular fracture surgery. J Orthop Trauma. 2013 Jan;27(1):11-5. doi: 10.1097/BOT.0b013e31824d96f6. PMID 22495529
- [Background] Manson TT, Nascone JW, Sciadini MF, O'Toole RV. Does fracture pattern predict death with lateral compression type 1 pelvic fractures? J Trauma. 2010 Oct;69(4):876-9. doi: 10.1097/TA.0b013e3181e785bf. PMID 20938275
- [Background] Manson TT, Nascone JW, O'Toole RV. Traction vertical shear pelvic ring fracture: a marker for severe arterial injury? A case report. J Orthop Trauma. 2010 Oct;24(10):e90-4. doi: 10.1097/BOT.0b013e3181dc2443. PMID 20871243